CLINICAL TRIAL: NCT01969045
Title: Effect of the EnkFiberoptic Atomizer Set on Usage of Anaesthetics During the Bronchoscopy
Acronym: EnkAtomizer
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: RWTH Aachen University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 13-103; EK 222/13 (Other: Ethics Committee University Hospital Aachen)
Record Dates: First submitted 2013-10-21; First posted 2013-10-24 (Estimated); Last update posted 2016-02-18 (Estimated); Status verified 2016-02

CONDITIONS: Administration of Local Anaesthetics With a Special Atomizing Set Durching Fexible Bronchoscopy
Keywords: felxible bronchoscopy; anaesthetics; transcutaneous pCO2; capillary pCO2
MeSH Terms: interventions — Bronchoscopes

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Working channel (Experimental): Patients will receive local anaesthetics via the working channel of the bronchoscope.
  Interventions: Device: bronchoscope
- Enk Fiberoptic Atomizer (Experimental): Patients will receive the local anaesthetics for the flexible bronchoscopy via the nebulizer Enk Fiberoptic Atomizer.
  Interventions: Device: Enk Fiberoptic Atomizer

INTERVENTIONS:
Device: Enk Fiberoptic Atomizer — Nebulization of local anesthetics with the Enk Fiberoptic Atomizer by Cook Medical during the felxible bronchoscopy
  Other Names: Enk Fiberoptic Atomizer Set, Cook Medical
  Arms: Enk Fiberoptic Atomizer
Device: bronchoscope — Standard procedure: Administration of local anesthetics via the working channel of the bronchoscope during the felxible bronchoscopy
  Arms: Working channel

SUMMARY:
The aim of this prospective study is to examine the benefits und risks of administration of local anaesthetics with a special atomizing set (Enk Fiberoptic Atomizer, Cook Medical) during flexible bronchoscopy.

ELIGIBILITY:
Inclusion Criteria:

* bronchoscopy with transbronchial biopsy or cryobiopsy indicated for diagnostic purposes (suspected lung cancer, interstitial lung disease, unexplained pulmonary opacities)
* hospitalized patients
* patients aged 18 years or above
* written informed consent prior to study participation

Exclusion Criteria:

* known allergy to local anesthetics, midazolam or propofol, known epilepsy, known severe neurological or psychiatric disorder, hemodynamic instability with need for vasopressor therapy, acute or chronic decompensated heart failure, respiratory failure with the need for oxygen supplementation of more than 2 l per minute at rest (pO2 > 55 mmHg) or pCO2 > 50 mmHg at ambient air, known upper airway anomalies, surgery or irradiation of the upper airways in the past, contraindication for transbronchial biopsy as published by international guidelines, e. g. bleeding disorders or severe pulmonary hypertension
* women, who are pregnant or breastfeeding
* alcohol or drug abuse
* expected non-compliance
* patients unwilling or unable to give informed consent, patients with limited ability to comply with instructions for this study
* Participation on another clinical trial within the last 3 months
* subjects who are committed to an institution and/or penitentiary by judicial or official order.
* employees of the investigator cooperation companies.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2014-02; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Amount of anaesthetics during fexible bronchoscopy | one hour
  Valdiation of the total amount of administered propofol (mg) during the fexible bronchoscopy.
  Usage of sedatives other than propofol (midazolam), total amount of administered lidocaine, duration of bronchoscopy.

SECONDARY OUTCOMES:
pCO2 | two hours
  Determination of:
  maximum transcutaneous pCO2 during bronchoscopy, mean transcutaneous pCO2 during bronchoscopy, capillary pCO2 immediately after bronchoscopy and 2 hours later, time to Aldrete Score of at least 9 after procedure

CONTACTS AND LOCATIONS:
Overall Officials: Tobias Müller, Dr. med., Principal Investigator — Department of Cardiology, Pneumology, Vascular Medicine and Intensive Care Medicine, RWTH Aachen University Hospital
Locations (1):
- Department of Cardiology, Pneumology, Vascular Medicine and Intensive Care Medicine, RWTH Aachen University Hospital, Aachen, North Rhine-Westphalia, Germany